CLINICAL TRIAL: NCT04417049
Title: Pentoxifylline for Bipolar Depression: A Proof-of-Concept Feasibility Study
Brief Title: Treatment of Bipolar Depression With Pentoxifylline
Acronym: PTX-BD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Joshua Rosenblat, Principal Investigator, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-5219
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Pentoxifylline

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pentoxifylline (Experimental)
  Interventions: Drug: Pentoxifylline 400 MG

INTERVENTIONS:
Drug: Pentoxifylline 400 MG — All patients will be provided with pentoxifylline 400 mg to be orally ingested twice daily for 8 weeks.
  Other Names: Trental

SUMMARY:
Growing theoretical and clinical evidence has suggested that pentoxifylline may have an effect in improving depressive symptoms. Herein, we aim to evaluate the effect of pentoxifylline in patients with bipolar depression over an 8-week trial.

DETAILED DESCRIPTION:
Growing evidence has demonstrated that inflammation and alterations in cerebral blood flow (CBF) contribute to the pathophysiology of bipolar depression (BD). Pentoxifylline is a phosphodiesterase inhibitor that improves CBF and has potent anti-inflammatory and antioxidant effects. We therefore hypothesize that pentoxifylline may have antidepressant effects in BD. We will conduct an 8-week, open-label, single-armed, feasibility study assessing clinical and neurobiological effects of adjunctive pentoxifylline in the acute treatment of BD. Feasibility will be determined by evaluating recruitment/retention rates, target engagement (e.g., changes in biomarkers with pentoxifylline treatment) and preliminary efficacy testing with 6 participants. Evaluating pentoxifylline's effects may further our understanding of BD pathophysiology and help identify novel treatment targets.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written, voluntary informed consent prior to study enrollment. Substitute decision makers will not be allowed to consent to study on a potential patients behalf.
2. Male or female between the age of 18 to 65, inclusive.
3. Meets DSM-5 criteria for Bipolar I or II Disorder, currently experiencing a Major Depressive Episode. Diagnosis will be confirmed using the Mini-International Neuropsychiatric Interview (MINI) conducted by a delegated physician or trained research study while assessing eligibility.
4. Patient must present with a moderate to severe depressive episode, as determined by the MADRS score greater than 21.
5. Patient must be receiving guideline-concordant pharmacotherapy without changes in the last month.

Exclusion Criteria:

1. Currently exhibiting symptoms of mania, as determined by the Young Mania Rating Scale (YMRS) score greater than 11.
2. Current symptoms of psychosis or perceptual disturbances of any kind per investigator discretion
3. History of neurological disorders
4. Presence of active suicidality, as determined by the MADRS suicidality item (Item #10) score greater than 4
5. Presence of a contraindication to PTX, including a drug allergy or allergy to xanthine derivatives, low or labile blood pressure, acute myocardial infarction, cardiac arrhythmia, peptic ulcers, coronary artery disease or coagulation disorder.
6. Renal impairment, assessed as creatinine clearance less than 80ml/min
7. Abnormal liver function, assessed as ALT or AST ≥ 3 x ULN or bilirubin ≥ 2 x ULN
8. Severe myocardial infarction
9. Patients with standard contraindications to magnetic resonance imaging (MRI), such as non-MRI compatible implanted metallic devices
10. Patients with a history of cerebrovascular disease or history of intercranial hemorrhage.
11. Laboratory biochemical evidence of abnormal bleeding and/or coagulopathy
12. Pregnant or breastfeeding women. Patients who are sexually active must agree to use a highly effective contraceptive method
13. Use of prohibited concomitant medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
The recruitment rate | 8 weeks
  The feasibility of pentoxifylline as a treatment in bipolar disorder will be measured by recruitment rate
The retention rate | 8 weeks
  The feasibility of pentoxifylline as a treatment in bipolar disorder will be measured by retention rate of the study.

SECONDARY OUTCOMES:
Safety will be assessed using patient-reported treatment emergent adverse events. | 8 weeks
Change in depression severity using the Montgomery Asberg Depression Rating Scale (MADRS) | 8 weeks
  The MADRS is a clinician-rated scale measuring depression severity. It consists of 10 items, each scored from 0 (normal) to 6 (severe), for a total possible score of 60. A higher score is indicative of greater depressive severity Response rates are defined as ≥ 50% decrease and Remission ≤ 10 actual score.
Change in cerebral blood flow using ASL MRI imaging | 8 weeks
  Patients will complete an MRI sequence called arterial spin labelling (ASL) at baseline and week 8 to look at changes in cerebral blood flow before and after treatment. ASL does not use any contrast or radiation.
Change in inflammatory markers using blood serum and plasma | 8 weeks
  Blood will be collected in order to evaluate changes in inflammatory biomarkers associated with depressive disorders (e.g., TNF-alpha, IL-1 and IL-6).
Change in subjective measures of depression using 16-item Quick Inventory for Depressive Symptomology-Self Report (QIDS-SR16) Total Score | 8 weeks
  Patients will complete a brief self-reported scale that measures subjective symptoms of depression. In total there are 16 items, each scored from 0 to 3. The total score ranges from 0 to 27, with higher scores indicating worse depressive severity.
Changes in subjective measures of cognition using the Perceived Deficits Questionnaire for Depression-5 item (PDQ-5-D) | 8 weeks
  The PDQ-5 is a brief patient-rated scale to assess subjective cognitive dysfunction in people with depression. The PDQ originally is a 20-item questionnaire that generates a total score and 4 subscale scores in 4 cognitive domains: attention/concentration, retrospective memory, prospective memory, and planning/organization. The 5-item version (PDQ-D-5) is derived from the 20-item version and provides a validated measure of perceived cognitive deficits in depressive disorders.
Changes in psychomotor speed, concentration and memory using the Digit Symbols Substitution Task (DSST) | 8 weeks
  The DSST is used to evaluate psychomotor speed and concentration. It consists of multiple digits with unique symbols associated with each digit. Patients are asked to substitute each digit with the correct symbol in 90 seconds. Each correct symbol is counted to calculate the total score
Change in attention and concentration using the Trails Making Tests | 8 weeks
  Trail Making Test (TMT) is a cognitive test designed to assess attention and concentration through visuomotor tracking, executive function, and cognitive flexibility. It consists of two parts, A and B. In part A, a line is drawn between consecutive numbers. In part B a line is drawn alternating between numbers and letters. Score is calculated through total time to completion of each part, with higher times indicating impairment.
Change in verbal fluency using the FAS test | 8 weeks
  Change in verbal fluency (i.e., semantic and animal naming) will be measured by using the Controlled Oral Word Association Test. Scores will be assessed through the total number of words stated in a given letter or category in a time period of one minute. Number of repetitions and intrusions will also be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Rosenblat, MD, MSc, Principal Investigator — Psychiatry
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No